CLINICAL TRIAL: NCT01342302
Title: An Online Psychoeducational Intervention for Young Women With Breast Cancer and Their Partners
Acronym: OPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Karen Fergus, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 200-2008
Record Dates: First submitted 2009-10-15; First posted 2011-04-27 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2011-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Couples; Distress; Online Support; e-health; Intervention; Relationships
MeSH Terms: conditions — Breast Neoplasms | interventions — Psychosocial Intervention; Family Characteristics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Couples Intervention (Other): Single arm study design
  Interventions: Behavioral: Psychosocial Intervention for Couples

INTERVENTIONS:
Behavioral: Psychosocial Intervention for Couples — Intervention delivered on line

SUMMARY:
Breast cancer is distressing for couples in general but even more so when the illness strikes at a relatively young age. In addition to common relationship challenges, younger couples have to contend with the loss or disruption of age-appropriate goals for themselves. Presently, there are virtually no resources designed specifically to assist young couples coping with breast cancer. The purpose of this study is to develop and evaluate an online educational program geared to the unique needs and demanding schedules of young couples. The purpose of the program is to improve couples' relationships and mutual coping. Seventeen couples will take part in the 7-week program. They will complete questionnaires before and after participating to evaluate the program's helpfulness. This study will allow for the creation of a user-friendly, cost-effective tool that could help to improve the lives of all young couples coping with breast cancer in the years to come.

DETAILED DESCRIPTION:
Women diagnosed with breast cancer at or before the age of 40 experience greater distress and poorer quality of life than women diagnosed later in life. In addition to having to cope with the range of issues common to all women with breast cancer, young women face unique challenges such as loss of fertility, concerns for young children, and interruptions to early-stage careers. The presence of adequate social support is a mitigating factor for distress in young women, and spousal support in particular has been shown to play a crucial and distinctive role in determining how well a woman adjusts to breast cancer. Unfortunately, the evidence suggests well-spouses are significantly distressed themselves, and often fall short in their attempts to meet the needs of their ill partners despite generally good intentions. Consequently, researchers have recommended that psychosocial interventions be geared to couples. However, traditional counseling interventions may not appeal to younger couples with numerous responsibilities and time constraints.

The purpose of this study is to examine the feasibility, process, and outcomes of an innovative online intervention tailored to the unique needs of young women and their partners. The primary goal is to improve partners' relationship functioning and capacity to work together as a team in relation to the illness. The secondary goal is to combat feelings of isolation by creating a community of similarly affected couples. The intervention will be delivered via a professionally moderated, password-protected website and entail: Information relevant to young couples with breast cancer; structured, interactive learning modules; and a discussion board. The online modality is particularly suited to the younger demographic targeted by this project because of its familiarity, comfort, convenience, and flexibility.

A non-randomized, repeated measures analysis of variance design will be used to test the intervention. Seventeen couples will be recruited within the Greater Toronto Area. Questionnaires assessing relationship functioning, psychological adjustment, and quality of life will be administered to participants at baseline and at completion of the 7-week program. Qualitative data from the website and treatment satisfaction questionnaire will be analyzed thematically in order to improve the intervention and its delivery.

The potential for this online intervention to fill a void in support options available to both young women with breast cancer and their partners is vast. Following completion of the project, not only will there be a demonstrable product in the website, but the investigators will have the knowledge with which to further test the intervention in a RCT. The ultimate impact of the proposed project will be the creation of an accessible, cost-effective, empirically validated tool that could help to improve the quality of life of all young couples coping with breast cancer, regardless of geographic location, in the years to come.

ELIGIBILITY:
Inclusion Criteria:

* woman has received a diagnosis of breast carcinoma within the last 18 months at any point in her treatment trajectory.
* Women must be free of known local recurrence or metastatic disease at the time of enrolment.
* Patients will have been 40 years of age or younger when diagnosed.
* Partners must be 45 years of age or younger at the time of diagnosis. - Couples must be heterosexual, and married, cohabitating, or engaged. - Participants must be fluent in English with the ability to read and write in English.
* All participants will require convenient access to a computer with internet connection.

Exclusion Criteria:

* All participants will be screened for mental illness that would interfere with their capacity to benefit from the program (e.g., suicidality, psychotic disorders, substance abuse) and excluded on this basis.
* Couples who plan to participate in couple or individual counselling during the 7-week study duration will be excluded.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in Dyadic Adjustment Scale (DAS) scores from pre (0 weeks) to post-treatment (7 weeks) | pre-treatment (0 weeks) and immediate post-treatment (7 weeks)
  The DAS assesses couple's level of relationship satisfaction. The DAS will be used to assess change in couples' level of relationship satisfaction following participation in the Couplelinks program over a 7 week period, from pre-treatment (0 weeks) to post-treatment (7 weeks).
Change in Personal Assessment of Intimacy in Relationships scale scores from pre (0 weeks) to post-treatment (7 weeks) | pre-treatment (0 weeks) and immediate post-treatment (7 weeks)
  The Personal Assessment of Intimacy in Relationships scale assesses the degree of feelings of intimacy between partners. This primary outcome measure will be used to assess changes in the degree of the feelings of intimacy between partners following participation in the Couplelinks program over a 7 week period, from pre-treatment (0 weeks) to post-treatment (7 weeks).

SECONDARY OUTCOMES:
Mental Psychological Development Questionnaire (MPDQ) | Pre-treatment (0 weeks) and immediate post-treatment (12 weeks).
  The MPDQ assesses individual psychological adjustment.
Mental Health Inventory (MHI) | pre-treatment (0 weeks) and post-treatment (7 weeks)
  The MHI assesses individual psychological adjustment.
Hospital Anxiety and Depression Scale (HADS) | pre-treatment (0 weeks) and immediate post-treatment (7 weeks)
  The HADS assesses individual psychological adjustment.
Functional Assessment of Cancer Therapy-Breast (FACT-B) | pre-treatment (0 weeks) and immediate post-treatment (7 weeks
  The FACT-B assesses women's individual physical and psychological adjustment to breast cancer treatment.
Breast Cancer and Relationship Measure | pre-treatment (0 weeks) and immediate post-treatment (7 weeks
  This measure assesses the impact of breast cancer on couple mutuality.
Treatment Expectancy and Motivation Measure (TEMM) | pre-treatment (0 weeks)
  The TEMM assesses the degree to which individuals believe that the treatment will be helpful to them prior to starting the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Fergus, PhD, Principal Investigator — Toronto Sunnybrook Regional Cancer Centre; Debbie McLeod, PhD, RN, Study Director — Cancer Care Program, Nova Scotia Cancer Centre; Ellen Warner, MD, Study Director — Toronto Sunnybrook Regional Cancer Centre; Sandra Gardner, PhD, Study Director — Toronto Sunnybrook Regional Cancer Centre; Margaret Fitch, RN, Study Director — Toronto Sunnybrook Regional Cancer Centre; Barbara Fitzgerald, RN, Study Director — Princess Margaret Hospital, Canada; Leeat Granek, PhD, Study Director — Toronto Sunnybrook Regional Cancer Centre
Locations (1):
- Sunnybrook Odette Cancer Centre, Toronto, Ontario, Canada